CLINICAL TRIAL: NCT05090345
Title: Prospective Multi Center Study of Pediatric Cellular Therapy Patients at Risk for Endothelial Dysfunction, Sinusoidal Obstruction Syndrome and/or Multi-Organ Dysfunction Syndrome (MODS)
Brief Title: A Prospective Registry of Pediatric Cellular Therapy Patients at Risk for Endothelial Dysfunction, Sinusoidal Obstruction Syndrome and/or Multi-Organ Dysfunction Syndrome (MODS).
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00112697; NCI-2021-11324 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2021-10-12; First posted 2021-10-22 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Hematopoietic Cell Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biorepository trial of children and adolescents/young adults (AYA): undergoing hematopoietic cell transplantation (HCT) to assess the impact of endotheliopathies in the HCT setting as a contributor of significant morbidity and mortality.
  Interventions: Other: Biorepository Trial

INTERVENTIONS:
Other: Biorepository Trial — participating in this arm, peripheral blood specimen(s) will be obtained at 8 specified time-points.

SUMMARY:
This is a prospective international multi-center registry and biorepository trial of children and adolescents/young adults (AYA) undergoing hematopoietic cell transplantation (HCT) to assess the impact of endotheliopathies in the HCT setting as a contributor of significant morbidity and mortality.

DETAILED DESCRIPTION:
Primary:

* To evaluate the proportion of pediatric patients undergoing hematopoietic cell transplant (HCT) who develop endotheliopathies (SOS, TMA, DAH and IPS) and/or MODS within 100 days of such therapies.
* To evaluate the proportion of pediatric patients undergoing hematopoietic cell transplant (HCT) who experience abnormal levels of circulating angiogenic, vascular permeability and inflammatory factors within 100 days post HCT-CT in the setting of endotheliopathies.

Secondary/Exploratory Objective(s):

* To determine the impact of endotheliopathies in the HCT setting on the overall survival.
* To assess the efficacy of specific prophylaxis and treatment strategies directed at endotheliopathies (SOS, TMA, DAH and IPS) post-HCT among enrolled children on overall survival.
* To assess whether exposure to immunotherapies (CAR-T, PD-1 Inhibitors, bispecific T-cell engager (BiTE) antibodies and antibody drug conjugates) prior to HCT affects post-HCT outcomes (endotheliopathies and MODS).

ELIGIBILITY:
Inclusion Criteria:

* Children, adolescents and young adults (AYA) 0-26 years of age undergoing HSCT.
* Recipients of autologous and allogeneic HSCT.
* Any preparative regimen.

Exclusion Criteria:

* Any patient who does not consent/assent to participation.
* Any patient for whom 5 mL blood sample(s) drawn at specified intervals would pose any more than minimal risk, as defined by institutional guidelines and at discretion of treating physician will be ineligible for biorepository banking.

Ages: 0 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children, adolescents and young adults (AYA) 0-26 years of age undergoing HSCT.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2026-02-05 (Estimated); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of pediatric patients undergoing hematopoietic cell transplant (HCT) who develop endotheliopathies (SOS, TMA, DAH and IPS) and/or MODS within 100 days of such therapies. | through study completion, an average of 1 year
Proportion of pediatric patients undergoing (HCT) who experience abnormal levels of circulating angiogenic factors within 100 days post HCT-CT in the setting of endotheliopathies. | through study completion, an average of 1 year
Proportion of pediatric patients undergoing (HCT) who experience abnormal levels of vascular permeability within 100 days post HCT-CT in the setting of endotheliopathies. | through study completion, an average of 1 year
Proportion of pediatric patients undergoing (HCT) who experience abnormal levels of inflammatory factors within 100 days post HCT-CT in the setting of endotheliopathies. | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Overall survival. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kris Mahadeo, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - Duke University, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Duke University Medical Center — http://www.dukehealth.org